CLINICAL TRIAL: NCT01176955
Title: A Novel Method for Improving Acne Outcomes
Brief Title: A Novel Method to Improve Acne Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00008982
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-06

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne vulgaris; Adherence; Compliance; MEMS; Benzoyl peroxide
MeSH Terms: conditions — Acne Vulgaris; Patient Compliance | interventions — Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet survey (Experimental): Subjects will receive a weekly email link to complete an internet survey about their acne and use of the study medication.
  Interventions: Behavioral: Internet survey; Drug: Benzoyl peroxide 5% gel
- Control (Placebo Comparator): Subjects will receive standard-of-care treatment with the study medication, without internet surveys.
  Interventions: Drug: Benzoyl peroxide 5% gel

INTERVENTIONS:
Behavioral: Internet survey — A weekly email link will be generated to an internet survey which questions subjects about their acne severity, compliance with the study medication, and attitudes toward acne and the study medication.
  Arms: Internet survey
Drug: Benzoyl peroxide 5% gel — Topical benzoyl peroxide 5% gel, to be used once daily to the face.

SUMMARY:
This is an investigator-blinded, prospective study of 20 subjects aged 13 through 18 with mild to moderate acne. Study subjects will be randomized to an internet survey group, in which an email link for a survey ascertaining the status of the subject's acne is sent weekly, or to a control group. All study subjects will use benzoyl peroxide 5% gel, and adherence and clinical improvement will be monitored over 12 weeks. The investigators hypothesis is that subjects in the internet survey group will have improved adherence to the study medication and clinical outcomes, because the weekly survey will remind subjects to use their medication.

ELIGIBILITY:
Inclusion Criteria:

* male or female 13 to 18 years of age with a diagnosis of mild to moderate acne vulgaris by a dermatologist.
* written consent of participation must be given by parent or guardian and child.

Exclusion Criteria:

* Age less than 13 or greater than 18 years of age.
* Known allergy or sensitivity to topical benzoyl peroxide gel in the subject.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication, topical or systemic, for acne vulgaris while participating in the study.
* Subjects may not use topical retinoids or other benzoyl peroxide products, including Proactiv® or topical prescription medications while enrolled in the study.
* Women that are actively trying to become pregnant or wish to become pregnant during the time frame the study is to take place will be excluded.
* Subjects will be carefully selected for this study and only those deemed appropriate for treatment with benzoyl peroxide will be placed on this medication.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Study Director — Wake Forest University
Locations (1):
- Wake Forest University Health Sciences, Department of Dermatology, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Subjects will receive standard-of-care treatment with the study medication, without internet surveys. Standard-of-care will mean patients are directed to take the medication daily and return for visits at 6 and 12 weeks.
Period: Overall Study
Arm/Group | Internet Survey | Control
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet Survey | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.49) | 15.5 (2.22) | 15.4 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Measured Adherence by the MEMS Cap in Relation to the Patient Reported Adherence Via the Internet Survey.
Description: Adherence will be objectively measured with the Medication Event Monitoring System (MEMS) cap and the percentage of prescribed doses taken will be reported. Study subjects' self-reported adherence (in the intervention group, via the weekly internet survey) will be compared to objectively measured adherence via MEMS caps. Adherence was monitored objectively with electronic monitors that recorded the date and time when the medication containers were opened (medication event monitoring system caps). Adherence was rated as a percentage of days the medication container was opened; adherence could be greater than 100% if the container was opened more than once per day.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: percentage of days containers were open
Arm/Group | Internet Survey | Control
Number analyzed (Participants) | 7 | 8
percentage of days containers were open | 74 [58 to 132] | 32 [4 to 80]

2. Secondary Outcome: The Change (Dynamic Assessment) in the Acne Global Assessment From Baseline to End of Study.
Description: Acne Global Assessment is measured by a study investigator and is an overall assessment of the subject's acne severity, on a 0 (clear) to 5 (very severe) scale.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Internet Survey: Patients received a weekly Internet survey to report on the status of their acne.
- Control: Patients received standard-of-care therapy without weekly Internet surveys.
Arm/Group | Internet Survey | Control
Number analyzed (Participants) | 7 | 8
units on a scale | -0.71 (0.76) | -0.25 (0.46)

3. Secondary Outcome: The Change (Dynamic Assessment) From Baseline to End of Treatment in Lesion Counts.
Description: Both inflammatory (papules, pustules and nodules) and non-inflammatory (open and closed comedones) acne lesions will be counted by a study investigator. Percentage change from baseline to the final study visit will be calculated.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Arm/Group | Internet Survey | Control
Number analyzed (Participants) | 7 | 8
percent change in lesion count | -36 (37) | -8 (65)

4. Secondary Outcome: The Measured Adherence by the MEMS Cap in Relation to the Change (Dynamic Assessment) in the Acne Global Assessment.
Description: All study subjects' objective adherence will be compared to clinical improvement as measured by the Acne Global Assessment.
Time Frame: 12 weeks
Measure: Number; unit: Spearman's Rank Correlation Coefficient
Groups:
- All Participants: This group includes all participants in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Spearman's Rank Correlation Coefficient | 0.53

ADVERSE EVENTS:
Arm/Group | Internet Survey | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No